CLINICAL TRIAL: NCT05641207
Title: A Clinical Evaluation of the RheOx Bronchial Rheoplasty System for the Treatment of the Symptoms of Chronic Bronchitis in Chinese Adult Patients With COPD
Brief Title: A Clinical Evaluation of the RheOx Bronchial Rheoplasty System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Energenx Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCS-001
Record Dates: First submitted 2022-11-17; First posted 2022-12-07 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Bronchitis; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: An intervention of a device product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental device RheOx™ with the RheOx™ Catheter was only used in the trial (Experimental): All of participants who signed the ICF and meet all of inclution and exclution criterias will be enrolled to experimental arm.
  Interventions: Device: RheOx™ with the RheOx™ Catheter treated in the trial

INTERVENTIONS:
Device: RheOx™ with the RheOx™ Catheter treated in the trial — Eligible patients be assigned two sessions of RheOx bronchial rheoplasty procedures
  * Treatment 1 is for the treatment of right lung
  * Treatment 2 is scheduled one month apart for left lung

SUMMARY:
This is a prospective, multicenter, single arm and open-label clinical trial to evaluate the performance, effectiveness and safety of RheOx™ system in the treatment of the symptoms of chronic bronchitis in adult moderate to severe COPD patients.

DETAILED DESCRIPTION:
Eligible patients will be assigned to two sessions of treatments with RheOx™ system.

Treatment 1, named initial procedure is scheduled at right lung. And then treatment 2 is planned to treat left lung one month apart from initial procedure.

Following-up post either RheOx procedure is scheduled at 2nd day discharged from hospital and day 14 (phone call) and 1 month.

Patients will undergo follow-up evaluations at Month 3, 6 and 12 post-treatment 2. And a phone call is also scheduled every two months post treatment 2 except the above.

The assessments will include quality of life questionnaires, pulmonary function testing, lung CT scan and monitoring any adverse events and also any changes in inhaled medication, unschedule clinic visit or ER visit and even hosptialization.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age is ≥35 years and ≤80 years
2. Subject has chronic bronchitis, defined as productive cough for three months in each of two successive years, whereas other causes of productive cough have been ruled out.
3. Subject has a CAT score ≥ 10.
4. Subject's responses to the first two questions of the CAT questionnaire sum to ≥ 7 points or the sum is 6 points and the subject's total CAT score is > 20 points.
5. Subject has a SGRQ score ≥ 25.
6. Subject has post -bronchodilator FEV1/FVC < 0.7.
7. Subject has post-bronchodilator FEV1 percent predicted of ≥ 30%.
8. Subject is receiving guideline directed pharmacotherapy which includes one or more long-acting bronchodilator (LAMA, LABA) with or without an inhaled corticosteroid for at least 8 weeks prior to enrollment.
9. Subject has a cigarette smoking history of at least ten pack years (packs per day x years of smoking), and has had quit smoking for at least 6 months before enrollment;
10. In the opinion of the investigator, subject is able to undergo 2 bronchoscopies under general anesthesia and is able to adhere to the study follow-up schedule.

Subject has provided informed consent.

Exclusion Criteria:

1. Subject has known unresolved lower respiratory tract infection (e.g., pneumonia, mycobacterium avium-intracellulare infection (MAI), fungus, tuberculosis).
2. Subject has a pulmonary nodule or cavity . In the judgement of the investigator, the subject may require intervention during the course of the study.
3. Subject has clinically significant bronchiectasis influencing the subject's clinical symptoms of cough and phlegm.
4. Subject has severe other lung diseases (including interstitial pneumonia, lung fibrosis, pulmonary fibrosis with emphysema, atelectasis, unresolved lung Cancer, giant pulmonary bullae);
5. Subject has asthma based on Global Initiative for Asthma (GINA) criteria.
6. Subject has had prior severe respiratory infection with SARS-CoV-2 (COVID-19) that required ICU support with non-invasive and/or invasive mechanical ventilation.
7. Subject had prior lung surgery, such as lung transplant, LVRS, lobectomy, lung implant/prosthesis, metal airway stent, valves, coils or bullectomy. Prior pneumothorax without lung resection, pleural procedures without surgery, or segmentectomy are acceptable
8. Subject has a history of arrhythmia within past two years which includes tachy-atrial arrhythmias, any ventricular tachy-arrhythmias, grade II, II or III AV transmission history of conduction blockor, sinus bradycardia with heart rate less than 45 beats per minute.
9. Subject is on anticoagulation for cardiovascular indications and, at the discretion of the investigator, is unable to have anticoagulants (i.e., Aspirin, Plavix, Coumadin) withheld for the bronchoscopy procedure per institution's standard of care.

   * If the anticoagulants withheld is clinically acceptable, five to seven days withheld before enrollment is advised.
10. Subject has other serious diseases (e.g. congestive heart failure, cardiomyopathy, or myocardial infarction in the past year, renal failure, liver failure, cerebrovascular accident within the past 6 months, uncontrolled diabetes (HbA1c >8%), uncontrolled hypertension (diastolic BP >100mmHg) or autoimmune disease requiring treatment with immunosuppressant medications or a disease requiring chemotherapy).
11. Subject has uncontrolled gastroesophageal reflux disease（GERD）that indicated by the common symptoms and signs like stomach burning, acid reflux, regurgitation of partial digested food or acid into throat.
12. Subject has any implantable electronic device (e.g., pacemaker, cardioverter defibrillator, neuro-stimulation devices).
13. Subject has known airway colonization with resistant organisms, such as pseudomonas, methicillin-resistant Staphylococcus aureus (MRSA), Burkholderia cepacia complex, Mycobacterium Tuberculosis (MTB), Mycobacterium abscessus mucor or significant fungus.
14. Subject has known severe pulmonary hypertension.
15. Subject has a known sensitivity to medication required to perform bronchoscopy (i.e., lidocaine, atropine, benzodiazepines, Propofol).
16. Subject has known allergy to nickel.
17. Subject is receiving any traditional Chines herbs for cough or phlegm. * mucolytics may be recommended by institute clinical practice, carbocysteine, oral or inhaled N-acetylcysteine, Eucalyptol and ambroxol hydrochloride are suggested.

    * The treatrment of this study is to ablate bronchial mucosa by airway intervention, then mucosa epithelium is repaired. The effect of inhalation on the repair of airway mucosal epithelium is unknown. Therefore, it is not recommended to oral or inhaled N-acetylcysteine during treatment and follow-up.
18. Subject has a steroid-dependent condition requiring >10 mg of oral corticosteroid (e.g. prednisone or equivalence.) per day.
19. Subject is unable to walk over 225 meters in 6 minutes.
20. Subject has emphysema of greater than or equal to 35% (low attenuation area≤ -950HU) as determined by HRCT quantitative analysis.
21. Subject is pregnant, nursing, or planning to get pregnant during study duration.
22. Subject has HIV infection or active syphilis infection;
23. Subject is currently participating in another clinical study involving an investigational product.
24. Subject is not suitable for bronchoscopy by the judgement of investigator.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-05-18 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) Score in Total | 6 Month after second RheOx procedure (treatment 2 on left lung )
  The mean change from baseline to Month 6. (The minimal is zero and maximal 40 points. The higher score means the impact is greater)

SECONDARY OUTCOMES:
CAT Score in Total | 12 months
  The mean change from baseline to 3，12 months (The minimal is zero and maximal 40 points. The higher score means the impact is greater)
St. George's Respiratory Questionnaire (SGRQ) | 12 months
  The mean change of SGRQ total score from baseline to 3，6 and 12 months(The minimal is zero and maximal 100 points. The higher score means the impact is greater)
CAT response rate | 12 months
  At 3, 6 and 12 months after RheOx procedures
SGRQ response rate | 12 months
  At 3, 6 and 12 months after RheOx procedures
Distal airway volume | Month 6
  The mean change from baseline to Month 6 in distal airway volume (DAV) at expiration, as determined by an independent core lab
Total Airway Counts | Month 6
  The mean change from baseline to Month 6 in Total Airway Counts(TAC) as determined by an independent core lab

OTHER OUTCOMES:
Cough and Sputum Questionnaire (CASA-Q) score | 12 months
  The mean change from baseline to 3, 6 and 12 months. (There are four dominants with its score range acordingly. Cough symptem 0-12, Cough Impact 0-32, Phlegm Symptem 0-12 and Phlegm Impact 0-24. The higher score indicates the better conditions)
Moderate and/or severe acute excerbation of COPD（AECOPD) post RheOx rheoplasty treatment | 12 months
  RheOx treatment to 12 months (30 days recovery period post treatment not included).
Total lung capacity(TLC), functional residual capacity (FRC) and inspiratory capacity (IC) | 6 months
  Change measured by computed tomograph scan at full breath-in and at end of tidal breath-out. Inspiratory capacity to be calculated by TLC minue FRC and the change from baseline to 6 months
6 minute walk distance(6MWT) | 12 months
  the mean change from baseline to 3, 6 and 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Guangfa WANG, MD, Principal Investigator — Peking University First Hospital
Locations (7):
- China (7):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Xinqiao Hospital, Army Medical University, Chongqing, Chongqing Municipality
  - First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Tenth People's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang